CLINICAL TRIAL: NCT03063125
Title: Perioperative Hypogonadism in Men Undergoing Radical Cystoprostatectomy for Bladder Cancer
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00140348
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Bladder Cancer; Low Testosterone Levels
Keywords: radical cystectomy; hypogonadism
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hypogonadism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bladder Cancer Patients: Patients with bladder cancer scheduled to undergo radical cystectomy (RC).

SUMMARY:
The purpose of this study is to examine the relationship between testosterone level changes around the time of radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bladder cancer
* Scheduled to undergo radical cystectomy

Exclusion Criteria:

* Evidence of advanced metastatic disease,
* Undergoing cystectomy for non-bladder primary malignancy or bladder cancer type other than urothelial cell
* History of breast or prostate cancer
* Polycythemia, cardiovascular thromboembolism, untreated obstructive sleep apnea, uncontrolled heart failure, or acute coronary event in the past six months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants are adult men undergoing RC for primary bladder cancer.
Study Population: Participants will be recruited from patients being treated at the University of Kansas Health System.Potiential patients will be recruited from the urology clinic, University of Kansas Cancer Center or during inpatient hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Holzbeierlein, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from University of Kansas Medical Center Urology Clinics
Period: Overall Study
Arm/Group | Bladder Cancer Patients
Started | 25
Completed | 23
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bladder Cancer Patients
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 18
Age, Continuous [Mean (Full Range); unit: years] | 68.9 [52 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Hypogonadism in Participants Based on Serum Testosterone 90 Days Post Radical
Description: The count of participants with hypogonadism (the level of serum testosterone used as a threshold).
Time Frame: 90 days post-RC surgery
Measure: Number; unit: participants
Arm/Group | Bladder Cancer Patients
Number analyzed (Participants) | 16
participants | 6

2. Secondary Outcome: The Number of Hypogonadism in Participants Based on Serum Testosterone 30 Days Post Radical Cystectomy
Description: The count of participants with hypogonadism 30 days post radical cystectomy using the serum testosterone levels (the level of serum testosterone used as a threshold).
Time Frame: 30 days post-RC surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bladder Cancer Patients
Number analyzed (Participants) | 11
Participants | 8

3. Secondary Outcome: The Number of Hypogonadism in Participants Based on Serum Testosterone Immediately Post Surgery Days Post Radical Cystectomy
Description: The count of participants with hypogonadism immediately post radical cystectomy based on levels of testosterone (the level of serum testosterone used as a threshold).
Time Frame: Immediately post-operatively RC surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bladder Cancer Patients
Number analyzed (Participants) | 20
Participants | 19

4. Secondary Outcome: The Number of Hypogonadism in Participants Based on Serum Testosterone at Baseline Days Post Radical Cystectomy
Description: The count of participants with hypogonadism at baseline days post radical cystectomy (the level of serum testosterone used as a threshold).
Time Frame: Baseline, prior to RC surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bladder Cancer Patients
Number analyzed (Participants) | 23
Participants | 12

ADVERSE EVENTS:
Time Frame: Patients were on trial for 3 months - this study was observational.
Description: Patients were on trial for 3 months - this study was observational.
Arm/Group | Bladder Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03063125/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT03063125/ICF_001.pdf